CLINICAL TRIAL: NCT04523116
Title: Validation of Tie2 as the First Tumour Vascular Response Biomarker for VEGF Inhibitors: Optimising the Design of a Subsequent Randomised Discontinuation Trial: VALTIVE1
Brief Title: Validation of Tie2 as the First Tumour Vascular Response Biomarker for VEGF Inhibitors: VALTIVE1
Acronym: VALTIVE1
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Manchester (Other)
Collaborators: Cancer Research UK (Other); Centre for Trials Research, Cardiff University (Unknown)
Responsible Party: Principal Investigator, Prof Gordon Jayson, Professor of Medical Oncology, University of Manchester
Other Study IDs: A29832
Record Dates: First submitted 2020-08-13; First posted 2020-08-21 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-10

CONDITIONS: Ovary Cancer
Keywords: VEGF inhibitors; Bevacizumab; Tie2; Biomarker; Ovarian
MeSH Terms: conditions — Ovarian Neoplasms; Venous Malformations, Multiple Cutaneous and Mucosal

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples will be collected from the participants twice before treatment with bevacizumab and once at the scheduled visits as per protocol.
  Blood will be separated at site through centrifugation and the plasma aspirated and separated into aliquots. These will be labelled and stored at a maximum of -20 C until they are shipped to the Christie NHS Foundation Trust Biochemistry Department.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Tumours require a blood supply to provide them with oxygen and nutrients and to enable spread of cancer through blood vessels to other organs (metastasis). The formation of new blood vessels is known as angiogenesis, which is controlled by a growth factor (like a hormone) called Vascular Endothelial Growth Factor (VEGF). Many drugs have been developed that block VEGF and, in most tumour types, including ovarian cancer, the addition of VEGF inhibitors (VEGFi) to conventional anti-cancer therapy postpones recurrence of the disease. In ovarian cancer, VEGFi improve the overall outcome from the cancer in patients who have advanced stage and high-risk disease. VEGFi are now widely used in cancer medicine, yet until now there have not been any biomarkers (tests) that could be used to tell patients and their doctors whether the drugs were working or not. This is important, as VEGFi have side effects that are unpleasant for the patient. Additionally, VEGFi treatments are expensive.

The VALTIVE team has discovered the first biomarker that informs doctors whether a VEGFi is blocking a tumour's blood supply. The test involves measuring a protein in the blood called Tie2, which can be measured from routine blood tests that patients have when going to the hospital. If the test shows that the amount of Tie2 decreases in the blood, it means that tumour blood vessels are blocked by VEGFi; if, on the contrary, the level increases, the blood vessels have escaped the control of VEGFi.

The investigators have shown that the Tie2 test works in their initial studies in ovarian and bowel cancer. In these studies, the Tie2 blood test was based in the research laboratories. The investigators now wish to establish the test in the Christie Hospital NHS Biochemistry laboratory in Manchester so that it can be used in clinical practice rather than just as a research tool. The investigators wish to measure the relationship between loss of control of VEGF inhibitors as measured by TIE 2 and other standard ways of measuring loss of control of the tumour like increases on CT scans. There are several reasons why this test is needed for patients with ovarian cancer:

* VEGFi are effective during a patient's first or subsequent treatments for advanced ovarian cancer, but it is not clear which individuals are benefitting from treatment whilst they are on treatment.
* Patients who have already had one course of VEGFi can be re-treated successfully.
* Patients can avoid needless side effects, if there is a way of demonstrating that the treatment is of no benefit to them.
* This test will help doctors choose the best drug to control ovarian cancer and how long to continue treatment. This is very important, since other maintenance therapies are now available and the optimal duration of VEGFi therapy is well known.
* Around the world many teams are developing new combination treatments including VEGFi. If these new combinations prove effective, it would be possible to use them as efficiently as possible, as they will be very expensive and may therefore be less accessible to patients.

These issues highlight the critical need to establish a test in the NHS that tells patients and their doctors when VEGFi are working and when they stop working.

In VALTIVE1 study, blood samples will be taken from patients who are receiving a VEGFi called bevacizumab for ovarian cancer. Patients' management will not change during their participation to the trial. The analysis of the blood sample will support the hypothesis that patients whose Tie2 level decreases in response to bevacizumab will have ovarian cancer that is controlled for much longer than those where the Tie2 level does not decrease. These results will be used to design a second trial where the investigators will prove conclusively the value of the Tie2 test.

The purpose of VALTIVE1 is to optimise sample acquisition time points and analytical algorithms to support the design of VALTIVE2, a randomised discontinuation trial. In VALTIVE2, Tie2-defined, vascular non-responding patients will be randomly allocated to stop bevacizumab after 9 weeks, by when a response can be detected, or to continue bevacizumab for the conventional year of treatment.

Both VALTIVE 1 and VALTIVE2 will test the theory that there is no advantage in continuing bevacizumab in a patient whose Tie2 level does not reduce in response to VEGFi.

DETAILED DESCRIPTION:
VALTIVE1 is a multi-centre, single arm, non-interventional biomarker study, which will enrol 176 participants who are 16 years or older and who have FIGO stage IIIc/ IV ovarian cancer on treatment with first-line platinum-based chemotherapy and bevacizumab. Potential participants will be identified at their treating hospital.

The definition of vascular response is either (i) stable or reduced concentrations of Tie2 after 6 weeks of treatment or (ii) a confirmed reduction in plasma Tie2 of >10% within 9 weeks of starting treatment.

Patients enrolled into the VALTIVE 1 study will provide blood samples twice before treatment with bevacizumab and then at the end Cycles 1, 2, and 3, at the end of cytotoxic chemotherapy, at 3 months, 6 months, 9 months, at the end of treatment, and at disease progression. The early samples will be used to refine the definition and number of required samples needed to define a Tie2-vascular response. Samples collected at 3 months, 6 months, 9 months, at the end of treatment, and at disease progression will be used to investigate the relationship between Tie2-defined vascular progression and RECIST1.1- or clinically-defined Progression Disease (PD).

While the patients receive single agent maintenance bevacizumab, patients will undergo RECIST1.1 scanning at 3 months, 6 months, 9 months, end of treatment and at disease progression, if not before. These scans will also be reported to RECIST 1.1.

Progressive disease will be defined by the date of radiological or clinically identified progressive disease or death.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible for participation in this trial, the patient must:

1. Be willing and able to provide written informed consent for the trial
2. Age 16 years or over on day of signing informed consent
3. 3. Histologically proven ovarian, primary peritoneal or fallopian tube cancer (henceforth referred to collectively as Ovarian Cancer - OC) FIGO stage III with residual disease of more than 1cm; or stage IV; or stage III at presentation treated with neoadjuvant chemotherapy; or stage III with contraindication to debulking surgery chemotherapy
4. Planned to receive treatment with bevacizumab or biosimilar bevacizumab
5. Be scheduled to receive at least 2 successive doses of bevacizumab with 6 or more weeks of follow up blood samples after the first dose of bevacizumab if given pre-operatively; or to start bevacizumab post-operatively
6. Be eligible for receiving treatment with first line, 3-weekly carboplatin and paclitaxel chemotherapy
7. Be willing to provide blood samples and comply with trial-specific procedures

Exclusion Criteria:

The patient must be excluded from participating in the trial if the patient:

1. Is unsuitable for treatment with VEGF inhibitors
2. Is unable or unwilling to comply with study procedures
3. Is participating in a clinical study with an investigational product other than carboplatin, paclitaxel and bevacizumab
4. Is judged by the investigator to be unlikely to comply with study procedures
5. Is pregnant or could become pregnant and is not using adequate contraception
6. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies)
7. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g. HCV RNA is detected). Testing only required if patient has a history of either of these

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Eligible participants are female patients with histologically proven Ovarian Cancer (OC) FIGO stage III.
Study Population: Potential participants will be under the care of a consultant who specialises in the treatment of ovarian cancer.
  Patients who have been diagnosed with stage III/IV ovarian cancer within the routine clinics of participating centres and identified as requiring treatment with bevacizumab will be approached and screened.
Sampling Method: Non-Probability Sample
Enrollment: 176 (Estimated)
Dates: Start 2021-01-14 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | Up to 12 months after completion of the last Participant's follow up visit
  To establish the validity of the Tie2 test as measured by progression free survival by showing the difference in terms of PFS between Tie2 vascular responders and Tie2 vascular non- responders.

SECONDARY OUTCOMES:
Definition of Tie2 defined vascular response Definition of Tie2 defined vascular response Definition of Tie2 defined vascular response Definition of Tie2 defined vascular response | Up to 12 months after completion of the last Participant's follow up visit
  To optimise the definition of Tie2-defined vascular response by analysing its relation with progression free survival as measured according to Response Evaluation Criteria in Solid Tumors(RECIST) v1.1 criteria.
Optimum number of blood samples | Up to 12 months after completion of the last Participant's follow up visit
  To define the optimum number of blood samples that need to be taken and tested for informing doctors whether their patients are responding to treatment (low level of Tie2) or are likely to progress (high level of Tie2).
Relation between surgery and Tie2 | Up to 12 months after completion of the last Participant's follow up visit
  Patients with advanced ovarian cancer have surgery which stimulates the formation of new blood vessels and, consequently, may increase the level of Tie2 in the blood. The measurement of Tie level in blood samples to be taken from 2 weeks before surgery until 4 weeks after surgery will show whether the surgery has any impact on plasma Tie2 concentrations.
Design of the subsequent trial, VALTIVE2 | Up to 12 months after completion of the last Participant's follow up visit
  The definition of vascular response as assessed by measurement of Tie2 levels in plasma and its relation with PFS as per RECIST criteria will be validated in the randomised discontinuation non-inferiority trial VALTIVE2.

CONTACTS AND LOCATIONS:
Overall Officials: Gordon Jayson, PhD, FRCP, Principal Investigator — University of Manchester
Locations (4):
- United Kingdom (4):
  - Royal United Hospitals Bath NHS Foundation Trust, Bath
  - The Christie NHS Foundation Trust, Manchester
  - East and North Hertfordshire NHS Trust, Northwood
  - University Hospital Southampton NHS Foundation Trust, Southampton

REFERENCES:
- [Derived] Holland-Hart D, Carucci M, Slusarczyk M, Longo M, Campbell S, Irving A, Noble S, Jayson G, Hopewell-Kelly N. Participants' perspectives of the advanced ovarian cancer biomarker study VALTIVE1: a qualitative study. BMJ Open. 2025 Jul 13;15(7):e088474. doi: 10.1136/bmjopen-2024-088474. PMID 40659403
- [Derived] Carucci M, Clamp A, Zhou C, Hurt C, Glasspool R, Monaghan PJ, Thirkettle S, Wheatley M, Mahmood M, Narasimham M, Cox T, Morrison H, Campbell S, Nelson A, Holland-Hart D, Hopewell-Kelly N, Thomas A, Porter C, Slusarczyk M, Irving A, Dive C, Adams R, Jayson GC. The VALTIVE1 study protocol: a study for the validation of Tie2 as the first tumour vascular response biomarker for VEGF inhibitors. BMC Cancer. 2024 Oct 24;24(1):1309. doi: 10.1186/s12885-024-13073-0. PMID 39448911